CLINICAL TRIAL: NCT05984485
Title: TME vs TME+nCT in Low-risk LARC
Brief Title: The Efficacy of Primary Total Mesorectal Excision (TME) Surgery Versus Neoadjuvant Chemotherapy Combined With TME Surgery in Low-risk Locally Advanced Rectal Cancer
Acronym: TaLaR-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-TaLaR-02
Record Dates: First submitted 2023-07-21; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; total mesorectal excision; neoadjuvant chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: 1. Primary TME
  2. neoadjuvant chemotherapy plus TME
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary total mesorectal excision (Experimental): Patients with low-risk locally advanced rectal cancer received total mesorectal excision alone.
  Interventions: Procedure: total mesorectal excision
- Neoadjuvant chemotherapy plus TME (Active Comparator): Patients with low-risk locally advanced rectal cancer received neoadjuvant chemotherapy and total mesorectal excision.
  Interventions: Procedure: neoadjuvant chemotherapy plus total mesorectal excision

INTERVENTIONS:
Procedure: neoadjuvant chemotherapy plus total mesorectal excision — Neoadjuvant chemotherapy regimen recommended FOLFOX6, XELON, FOLFOX, mFOLFOX for 4-6 courses, and TME surgical treatment after preoperative tumor restaging 1-2 weeks after neoadjuvant chemotherapy.
  Arms: Neoadjuvant chemotherapy plus TME
Procedure: total mesorectal excision — Standard total mesorectal excision
  Arms: Primary total mesorectal excision

SUMMARY:
Comparative analysis of the clinical efficacy between primary Total Mesorectal Excision (TME) surgery and neoadjuvant chemotherapy combined with TME surgery for low-risk locally advanced rectal cancer. Randomly enrolling eligible patients into either the control group receiving neoadjuvant chemotherapy combined with TME surgery or the experimental group receiving primary TME surgery, and subsequently comparing the clinical outcomes of the two groups

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients, aged 18 to 75 years;
2. Pathologically confirmed rectal adenocarcinoma;
3. Distance of the lower margin of the rectal tumor lesion from the anal margin <15cm;
4. High-resolution MRI indicates low-risk locally advanced rectal cancer: T1-3bN1-2 or T3aN0 or T3bN0; no involvement of the anal sphincter; negative mesorectal fascia (MRF) status; negative extramural vascular invasion (EMVI); no cancer nodules;
5. Exclusion of patients with non-local recurrence or distant metastases;
6. Absence of synchronous colorectal multiple primary cancers;
7. Adequate physical condition to tolerate surgery and neoadjuvant chemotherapy, including cardiac, pulmonary, hepatic, and renal functions;
8. The study physician assessed no difficulty in sphincter preservation;
9. patients and their families will be willing to participate in this study and provide written informed consent.

Exclusion Criteria:

1. Patients with concurrent other malignancies or a history of malignant tumors in the past;
2. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, or other conditions requiring emergency surgery;
3. Patients with tumor invasion into the external sphincter or levator ani muscles, or involvement of adjacent organs necessitating combined organ resection;
4. Patients with poor anal function or fecal incontinence before surgery;
5. Patients with a history of inflammatory bowel disease or familial adenomatous polyposis;
6. Patients recently diagnosed with other malignancies;
7. Patients with ASA grade ≥ IV and/or ECOG performance status score > 2;
8. Patients with severe liver or kidney dysfunction, significant cardiopulmonary impairment, coagulation disorders, or those with extreme underlying conditions unable to tolerate surgery;
9. Patients with a history of severe mental illness;
10. Pregnant or lactating women;
11. Patients with uncontrolled infections before surgery;
12. Patients with other clinical or laboratory conditions, as determined by the investigator, that render them unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
3-year Disease Free Survival | 3 years after surgery
  Defined as the proportion of patients who did not experience any of the following events from the beginning of the randomized subgroup to the end of the third year, which included disease progression, local recurrence, distant metastasis, or second primary colorectal cancer, or death from any cause.

SECONDARY OUTCOMES:
Distance from the inferior resection margin to the tumor | Immediately after the surgery
  The length between inferior resection margin and the tumor.
The status of circumferential margin | Immediately after the surgery
  When the distance from the tumor or malignant lymph node to the circumferential margin was ≤ 1 mm, it was recorded as a positive circumferential margin.
The status of distal resection margin | Immediately after the surgery
  When the distance from the tumor to the distal resection margin was ≤ 10 mm, it was recorded as a positive distal resection margin.
Postiveoperative stay | 1 months after surgery
  The days after surgery in the hospital
Time to Postoperative first feed | 1 months after surgery
  The duration after surgery to first feed
Time to Postoperative first gas | 1 months after surgery
  The duration after surgery to first gas
Postoperative pain | 1 months after surgery
  Postoperative pain according to pain socres
Postoperative anal function | 3 years after the surgery
  Anal function would be based on wexner Incontinence score. A total score of less than ten is considered good, and a score of more than ten is considered poor.
Quality of life score | 3 years after the surgery
  Quality of life score would be based on EORTC QoL C30 scale.
3-year overall survival | 3 years after the surgery
5-year Disease Free Survival | 5 years after the surgery
5-year overall survival | 5 years after the surgery
Number of participants with treatment-related adverse events | 1 month after neoadjuvant chemotherapy
  It would be assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Liang Kang, PhD,MD, Principal Investigator — Sun yat-sen University, sixth affiliated hospital
Locations (6):
- China (6):
  - Daping Hospital, Amy Medeical Univerisity, Chongqing, Chongqing Municipality
  - Sun yat-sen University, the Sixth Affiliated Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Nanchong Central Hospital of North Sichuan Medical College, Nanchong, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests can provide relevant data, but must be used anonymously